CLINICAL TRIAL: NCT04149626
Title: Prospective, Randomized Comparative Study of Intravenous Dexmedetomidine for Sedation in Orthopedic Surgery Under Regional Anesthesia
Brief Title: Dexmedetomidine Sedation in Orthopedic Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Collaborators: Maria Tileli (Unknown); Chryssoula Staikou (Unknown)
Responsible Party: Principal Investigator, Alexandros Makris, Consultant Anesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14720/29-10-2019
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Hallux Valgus and Bunion; Sedation
MeSH Terms: conditions — Hallux Valgus; Bunion | interventions — Dexmedetomidine; Midazolam; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Dexmedetomidine sedation
  Interventions: Drug: Dexmedetomidine
- Group B (Active Comparator): Midazolam sedation
  Interventions: Drug: Midazolam
- Group C (Active Comparator): Remifentanil sedation
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Sedation using dexmedetomidine (initial bolus dose followed by continuous infusion)
  Arms: Group A
Drug: Midazolam — Sedation using midazolam (initial bolus dose followed by continuous infusion)
  Arms: Group B
Drug: Remifentanil — Sedation using remifentanil (initial bolus dose followed by continuous infusion)
  Arms: Group C

SUMMARY:
60 patients ASA I-III, undergoing orthopedic surgery will be randomly assigned into one of three groups, namely group A (n=20), where dexmedetomidine will be used for sedation (initial bolus dose followed by continuous infusion), group B (n=20) where midazolam will be used for sedation (initial bolus dose followed by continuous infusion) and group C (n=20), where remifentanil will be used for sedation (initial bolus dose followed by continuous infusion). All patients will receive spinal anesthesia. Duration of postoperative analgesia, total dose of patient controlled IV morphine, sedation scores, nausea and vomiting, time of ambulation, sleep quality and patient satisfaction will be recorded for the first postoperative day. Additionally chronic pain on the site of surgery will be recorded in 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Physical status according to American Society of Anesthesiologists (ASA) I-III Patients scheduled for orthopedic surgery

Exclusion Criteria:

Patient denial, contraindication of spinal anesthesia or any of the agents used in the protocol, BMI above 30, Serious psychiatric, mental and cognitive disorders, Language barrier, illicit substances abuse,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia duration | 24 hours
  Time of first demand for analgesia (PCA first bolus dose)

SECONDARY OUTCOMES:
Postoperative pain: Numerical Rating Scale (NRS) | 24 hours
  Numerical Rating Scale (NRS) scores (Range 0-10, 0=no pain, 10=the worse pain ever)
Morphine consumption | 24 hours
  Doses requested, morphine consumption in mg
Rescue analgesia | 24 hours
  Paracetamol in mg consumed
Sedation | 24 hours
  Ramsay Sedation Scale (numeric score from 1 to 6, based on responsiveness of the patient)
Complications | 24 hours
Delirium occurence | 24 hours
  Nu-DESK scale (presence of disorientation, inappropriate behavior, inappropriate communication,illusions/hallucinations, psychomoter retardation). Each of the 5 items is rated from 0 to 2. A total of 10 is the maximum score. A score of more than 2 identifies the presence of delirium.
Chronic pain: Graded Chronic Pain Scale (GCPS) | 6 months
  Using of Graded Chronic Pain Scale (GCPS) Grade 0: No pain in prior 6 months Grade 1: Low Intensity - Low Disability Grade II: High Intensity Characteristic Pain Intensity - Low Disability Grade III: High Disability - Moderately Limiting Grade IV: High Disability - Severely Limiting

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Greece

IPD SHARING:
Plan to Share IPD: No